CLINICAL TRIAL: NCT01922544
Title: Conventional Versus EP-Catheter Guided Implantation of Coronary Sinus Lead in Patients Undergoing Cardiac Resynchronization Therapy
Brief Title: EP-Catheter Guided CS-Lead Implantation
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Fikret Er, Dr., University of Cologne
Other Study IDs: CRT1
Record Dates: First submitted 2013-08-11; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure; Reduced Left Ventricular Ejection Fraction; Left Bundle Branch Block
Keywords: heart failure; cardiac resynchronization therapy; coronary sinus lead
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Conventional group: In this group CS lead was implanted in a conventional manner.
- EP-catheter group: In this group coronary sinus was canulated using a steerable electrophysiology catheter.

SUMMARY:
In patients undergoing CRT device implantation a lead positioning in the coronary sinus is required. Even this part of the surgical procedure is challenging. In this study we compared retrospectively to methods of CS-lead implantation: conventional vs. EP-catheter guided.

ELIGIBILITY:
Inclusion Criteria:

* CRT implantation due to heart failure
* full documented data

Exclusion Criteria:

* previous pacemaker/ICD/CRT implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic heart failure and reduced left ventricular ejection fraction. Asynchronic contraction of left and right ventricle was reflected by QRS duration > 120 ms in left precordial leads.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Total Fluoroscopy Time | During implantation
  During CRT device implantation fluoroscopy is used and the total fluoroscopy time is counted.
Contrast medium account | During surgical procedure
  contrast medium is used and counted during crt device implantation.

SECONDARY OUTCOMES:
Successful implantation | During surgical procedure
  Successful crt implantation was defined as effective positioning of RV and CS lead +/- right atrial lead.

OTHER OUTCOMES:
Procedure related complications | 24 hours after start of surgery
  All complications during time frame of 24 hours after start of surgery were proved whether they were procedure related.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, Cologne, North Rhine-Westphalia, Germany